CLINICAL TRIAL: NCT02033239
Title: A Trial Investigating the Pharmacodynamic Response of FIAsp in Subjects With Type 1 Diabetes
Brief Title: A Trial Investigating the Pharmacodynamic Response of Faster Acting Insulin Aspart in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3887; 2011-001580-41 (EudraCT Number); U1111-1120-3772 (Other: WHO)
Record Dates: First submitted 2014-01-09; First posted 2014-01-10 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FIAsp (Experimental): Each subject will be randomised to a treatment sequence consisting of 8 treatment periods
  Interventions: Drug: Faster-acting insulin aspart
- NovoRapid® (Active Comparator): Each subject will be randomised to a treatment sequence consisting of 8 treatment periods
  Interventions: Drug: insulin aspart

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Subjects will receive different dose levels of faster acting insulin aspart and NovoRapid®. Single dose of trial products will be administered subcutaneously (s.c. under the skin).
  Arms: FIAsp
Drug: insulin aspart — Subjects will receive different dose levels of faster acting insulin aspart and NovoRapid®. Single dose of trial products will be administered subcutaneously (s.c. under the skin).
  Arms: NovoRapid®

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the pharmacodynamic (the effect of the investigated drug on the body) response of Faster acting insulin aspart (FIAsp) in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-64 years (both inclusive) at the time of signing informed consent
* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index 18.5-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking at least one cigarette, cigar or pipe daily)
* Not able or willing to refrain from smoking and use of nicotine substitute products during the inpatient period

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve | From 0 to 12 hours

SECONDARY OUTCOMES:
Area under the serum insulin aspart concentration-time curve | From 0 to 12 hours
Maximum glucose infusion rate | Within 0 to 12 hours after dosing
Maximum observed serum insulin aspart concentration | Within 0 to 12 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Background] Heise T, Stender-Petersen K, Hovelmann U, Jacobsen JB, Nosek L, Zijlstra E, Haahr H. Pharmacokinetic and Pharmacodynamic Properties of Faster-Acting Insulin Aspart versus Insulin Aspart Across a Clinically Relevant Dose Range in Subjects with Type 1 Diabetes Mellitus. Clin Pharmacokinet. 2017 Jun;56(6):649-660. doi: 10.1007/s40262-016-0473-5. PMID 27878566
- [Background] Heise T, Pieber TR, Danne T, Erichsen L, Haahr H. Faster Onset and Greater Early Exposure and Glucose-Lowering Effect with Faster-Acting Insulin Aspart vs. Insulin Aspart: A Pooled Analysis in Subjects with Type 1 Diabetes. Diabetes. 2016; Suppl. 1: A239. doi:10.2337/db16-861-1374 http://dx.doi.org/10.2337/db16-861-1374
- [Derived] Heise T, Pieber TR, Danne T, Erichsen L, Haahr H. A Pooled Analysis of Clinical Pharmacology Trials Investigating the Pharmacokinetic and Pharmacodynamic Characteristics of Fast-Acting Insulin Aspart in Adults with Type 1 Diabetes. Clin Pharmacokinet. 2017 May;56(5):551-559. doi: 10.1007/s40262-017-0514-8. PMID 28205039
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com